CLINICAL TRIAL: NCT06081790
Title: Simulated-based Training Program for Peripheral Nerve Blocks Under Ultrasound, in Anesthesia Residents: Learning Curve and Transference
Brief Title: Simulated-based Program for Peripheral Nerve Blocks in Anesthesia Residents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Pablo Miranda, MD, assistant professor, Pontificia Universidad Catolica de Chile
Other Study IDs: 230316005
Record Dates: First submitted 2023-09-14; First posted 2023-10-13 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Simulated - Based Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this Simulated Based Program for Peripheral Nerve Blocks is build learning curves in anesthesia residents.

The research questions are:

How behave the learning curves in a simulate based training program in peripheral nerve blocks in anesthesia residents? Does the learning achieved during the program transferred to the real patient's scenario?

Participants will be subjected to 10 simulated training sessions of a sciatic popliteal nerve block, subsequently their performance will be recorded and a global scale will be applied and movements will be measured. In a second stage, the same subjects will perform a block on a real patient to determine the transfer of this simulated learning.

ELIGIBILITY:
Inclusion Criteria:

- Anesthesia first year residents

Exclusion Criteria:

* Previous regional anesthesia rotation
* Previous training in ultrasound guided punction

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: First year Anesthesia Residents
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-04-04 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
observational global rating scale scores (GRS) | Pre-intervention: first measurement before simulated-based training. During intervention: We will assess participants after each training session during 10 weeks. Post intervention: measurement once finished the protocol. Up to 12 weeks
  At the end of the training, residents performance will be asses using a previous validated GRS (points 0-50)

SECONDARY OUTCOMES:
Total path length (TPL) | Pre-intervention: first measurement before simulated-based training. During intervention: We will assess participants after each training session during 10 weeks. Post intervention: measurement once finished the protocol. Up to 12 weeks
  At the end of the training, residents performance will be asses using a hands tracking motion device that measured TPL of both hand in meters

IPD SHARING:
Plan to Share IPD: No
After the end of the protocol the videos will be deleted

REFERENCES:
- [Result] Neal JM, Gerancher JC, Hebl JR, Ilfeld BM, McCartney CJ, Franco CD, Hogan QH. Upper extremity regional anesthesia: essentials of our current understanding, 2008. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):134-70. doi: 10.1097/AAP.0b013e31819624eb. PMID 19282714
- [Result] Hopkins PM. Does regional anaesthesia improve outcome? Br J Anaesth. 2015 Dec;115 Suppl 2:ii26-33. doi: 10.1093/bja/aev377. PMID 26658198
- [Result] Barrington MJ, Viero LP, Kluger R, Clarke AL, Ivanusic JJ, Wong DM. Determining the Learning Curve for Acquiring Core Sonographic Skills for Ultrasound-Guided Axillary Brachial Plexus Block. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):667-670. doi: 10.1097/AAP.0000000000000487. PMID 27685348
- [Result] Corvetto MA, Pedemonte JC, Varas D, Fuentes C, Altermatt FR. Simulation-based training program with deliberate practice for ultrasound-guided jugular central venous catheter placement. Acta Anaesthesiol Scand. 2017 Oct;61(9):1184-1191. doi: 10.1111/aas.12937. Epub 2017 Jul 6. PMID 28685812
- [Derived] Miranda PF, Araneda AL, Molina NP, Miranda FG, Morrison C, Corvetto MA, Altermatt FR. Simulated-based training for ultrasound-guided popliteal sciatic nerve block: determining the learning curve and transference to real patient. Adv Simul (Lond). 2025 Nov 11;10(1):55. doi: 10.1186/s41077-025-00389-5. PMID 41219804